CLINICAL TRIAL: NCT05039658
Title: A Phase Ib, Open Label, Randomized, Multicenter Study of the Efficacy and Safety of IBI110 Single Agent and in Combination With Sintilimab for Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma (r/r DLBCL)
Brief Title: Efficacy and Safety of IBI110 Single Agent and in Combination With Sintilimab in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma (r/r DLBCL)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI110B201
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: DLBCL
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single agent treatment arm with IBI110 (Experimental): IBI110 administered at RP2D
  Interventions: Drug: IBI110
- Combination treatment arm with IBI10 and sintilimab (Experimental): IBI110 and sintilimab administered at RP2D
  Interventions: Drug: IBI110 plus sintilimab

INTERVENTIONS:
Drug: IBI110 plus sintilimab — Sintilimab is a NMPA approved high-affinity, ligand-blocking, humanized anti-programmed death-1 (PD-1) IgG4 antibody that blocks the binding of Programmed death-ligand 1 (PD-L1) and programmed death-ligand 2 (PD-L2) to PD-1.
  Arms: Combination treatment arm with IBI10 and sintilimab
Drug: IBI110 — BI110 is a high-affinity, ligand-blocking, humanized anti- Lymphocyte Activation Gene-3 (LAG-3) IgG4 antibody that blocks the binding of LAG-3 to MHCII.
  Arms: Single agent treatment arm with IBI110

SUMMARY:
The purpose of this study is to determine whether treatment with IBI110 single agent and in combination with sintilimab demonstrates sufficient efficacy/safety in r/r DLBCL.

DETAILED DESCRIPTION:
This is a phase Ib, open-label, randomized study to determine the efficacy and safety of treatment with IBI110 single agent and in combination with sintilimab in DLBCL that are relapsed and/or refractory to available standard of care therapies.

Participants in each cohort are randomly assigned to one of the two arms: IBI110 single agent arm and IBI110 in combination with sintilimab arm. Participants received study treatment for a maximum of 2 years, or until disease progression (assessed by investigator per Lugano 2014 Criteria for Malignant Lymphoma (Cheson et al 2014)), unacceptable toxicity, death or discontinuation from study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18-70 years old (at the time consent is obtained)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Histologically confirmed diagnosis of DLBCL in a subject who has been pretreated with at least 2 lines of systematic treatment (regimens containing anthracyclines and anti-CD20 immunotherapy must be included);
* Subjects whose most recent therapy was CAR-T cell therapy were also eligible.

Exclusion Criteria:

Patients previously exposed to any anti-LAG-3 treatment.

* History of ≥Grade 3 CRS, neurotoxicity, or hemophagocytic lymphohistiocytosis) during previous CAR-T cell therapy.
* Impaired cardiac function or clinically significant cardiac disease.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease within two years prior to screening with a few exceptions as per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-27 (Estimated); Primary Completion 2022-07-12 (Estimated); Study Completion 2022-12-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  Percentage of subjects achieving complete remission and partial remission in the studied cohort
The frequency of adverse events (adverse events, AEs) and serious adverse events (SAEs) | Up to 24 months
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE were defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.

SECONDARY OUTCOMES:
complete response rate | Up to 24 months
  The percentage of subjects that achieved complete response in the studied cohort
DoR | Up to 24 months
  DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the the Lugano 2014 criteria or death regardless of cause.
PFS | Up to 24 months
  PFS is defined as the time from the treatment date to the date of disease progression per Lugano 2014 criteria or death regardless of cause.
OS | Up to 24 months
  OS is defined as the time from treatment to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No